CLINICAL TRIAL: NCT05560048
Title: Anti-exercise-fatigue Effects of Rice Protein RP-80NY in Men
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chung Shan Medical University (Other)
Collaborators: VEDAN Enterprise Corporation (Unknown)
Responsible Party: Principal Investigator, Chin-Lin Hsu, Professor, Chung Shan Medical University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: CS2-22067
Record Dates: First submitted 2022-09-16; First posted 2022-09-29 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment to placebo (Experimental): Participants should eat rice protein RP-80NY once a day for 28 days, then exchange the treatment sample to placebo after 14 days of wash-out. The dosage of the rice protein RP-80NY or placebo is 0.053 g/kg body weight.
  Interventions: Dietary Supplement: rice protein RP-80N; Dietary Supplement: placebo
- placebo to treatment (Experimental): Participants should eat placebo once a day for 28 days, then exchange the treatment sample to rice protein RP-80NY after 14 days of wash-out. The dosage of the rice protein RP-80NY or placebo is 0.053 g/kg body weight.
  Interventions: Dietary Supplement: rice protein RP-80N; Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: rice protein RP-80N — rice protein RP-80NY were dried beige powder. It can be stored at room temperature, but it must be exposed to direct sunlight
Dietary Supplement: placebo — placebo were dried beige powder. It can be stored at room temperature, but it must be exposed to direct sunlight

SUMMARY:
The aim of this study is to investigate the anti-exercise-fatigue effects of rice protein RP-80NY in men

DETAILED DESCRIPTION:
Each subject must undergo a maximum oxygen consumption test 1 week before the intervention (day 1), eat the test food for 28 days (day 1 to day 28), following 14 days of wash-out (day 29 to day 42), and undergo second maximum oxygen consumption test (day 43) and another test food intervention (day 43 to day 70). The assays of anthropometric measurement, diet questionnaire survey, grip strength test and fecal collection were carried out before and after the intervention (the 1st ,28th ,43th and 35th day). Each subject has to join the Wingate anaerobic test (day 21 and day 63), and the endurance exercise test (day 28 and day 70) during the intervention. All of the trial period was 70 days, and the blood samples of the subject will be collected at the times of exercise beginning, 15 min after exercise, the end of exercise, 1 hour after rest, 2 hour after rest ,and 3 hour after rest. During the whole period of participating in the program, blood will be collected 14 times, the blood volume of each times is 10 mL. Gas is collected before the period and within 1 hour, 2 hour and 3 hour after exercise (5 minute at a time). After intervention, the exercise time, oxygen intake, blood biochemical value and gut microbiota will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* The subject is a male and aged 20-40.
* The subject has a usual exercise habit (exercising 2 times or more per week) and did not participate in professional sports competitions or professional sports training during the study period.
* No smoking or drinking habits.
* No food allergies and the liver function is normal.
* No cardiovascular diseases or other chronic diseases, and no serious illnesses requiring hospitalization during the study period.
* The subject can understand the test process described in the consent form and the possible potential risks and benefits, and can sign the consent form.
* The subject can accept dietary control during the trial period.

Exclusion Criteria:

* Those who have taken nutritional supplements containing branched-chain amino acids.
* Those who cannot complete the wingate anaerobic test and the endurance exercise test.
* Those who are diagnosed with kidney disease, heart disease, or cancer and are still under active treatment.
* Have used other drugs, whose pharmacological effects may affect fatigue.
* Subjects who have systemic infections and require systemic antibiotics.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-09-30 (Actual); Primary Completion 2022-12-15 (Estimated); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
Change the exercise performance after intervention compare the exercise | 21th day, 63th day
  Duration of exhaustive exercise test (second) between pre- and post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Jou Chien, PhD student, Principal Investigator — Chung Shan Medical University; Ching-Fang Yang, MS student, Principal Investigator — Chung Shan Medical University
Locations (1):
- Chung Shan Medical University, Taichung, Taiwan